CLINICAL TRIAL: NCT06004180
Title: Interventional, Exploratory, Open-label Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Properties of Lu AF28996 in Japanese Men and Women With Parkinson's Disease
Brief Title: A Trial Investigating Lu AF28996 in Adult Japanese Participants With Parkinson's Disease (PD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20399A
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF28996 (Experimental): Participants will receive ascending oral doses of Lu AF28996 OD for 14 days (Day 1 to Day 14). From Day 15, the participant will initiate down-titration of Lu AF28996 as per investigator's judgement.
  Interventions: Drug: Lu AF28996

INTERVENTIONS:
Drug: Lu AF28996 — Hard capsule, orally, per schedule specified in the arm description.

SUMMARY:
This trial will evaluate the effects of Lu AF28996 in adult Japanese men and women with Parkinson's disease (PD). The main goals of the trial are to learn more about a) the safety and tolerability of Lu AF28996 (any new or worsening medical issues the participants have with treatment), and b) the pharmacokinetic parameters of Lu AF28996 (how the drug is absorbed, distributed, and processed by the body). Participants will take Lu AF28996 capsules orally once a day (OD). The participants will start with a low dose of Lu AF28996, which will be increased gradually over a period of 2 weeks, and then decreased gradually over a period of about 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant is diagnosed with idiopathic PD (consistent with the United Kingdom Parkinson's Disease Society Brain Bank Criteria for the Diagnosis of Parkinson's Disease) and should not have more than 1 first-degree relative with PD.
* The participant's Modified Hoehn and Yahr score is ≤3 in the ON state and ≤4 in the OFF state.
* The participant experiences well-recognizable and predictable motor fluctuations (≥1.5 hours of OFF-periods in the awake time, predictable morning OFF episodes included) causing clinically significant disability during the 7-week Screening Period.
* The participant currently has a good response to levodopa and has been receiving a stable dose of levodopa (≥3 doses per day of levodopa/dopa decarboxylase inhibitor therapy) ≥4 weeks prior to screening.
* The participant is Japanese, defined as having four Japanese grandparents and being born in Japan.

Exclusion Criteria:

* The participant has or had one or more of the following conditions that are considered clinically relevant in the context of the study; other neurological disorder, psychiatric disorder, seizure disorder or encephalopathy, respiratory disease, hepatic impairment or renal insufficiency, metabolic disorder, endocrinological disorder, hematological disorder, infectious disorder, any clinically significant immunological condition, or a history of narrow-angle glaucoma.
* The participant has a positive test result for SARS-CoV-2 at the Baseline Visit.
* The participant has undergone a neurosurgical intervention for PD (such as pallidotomy, thalamotomy, fetal or stem cell transplantation or deep brain stimulation).

Note: Other inclusion and exclusion criteria may apply.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From the day of first dose of study drug (Day 1) up to Day 35
Area Under the Plasma Concentration-Time Curve From Zero to Last Quantifiable Concentration (AUC0-tlast) of Lu AF28996 | Day 1 to Day 14 (0 [predose] to 15 hours postdose); Day 15 (24 hours post the Day 14 dose and before dosing on Day 15); and Day 16
Area Under the Plasma Concentration-Time Curve From Zero to 24 Hours Post-Dose (AUC0-24h) of Lu AF28996 | Day 1 to Day 14 (0 [predose] to 15 hours postdose); Day 15 (24 hours post the Day 14 dose and before dosing on Day 15); and Day 16
Maximum Observed Plasma Concentration (Cmax) of Lu AF28996 | Day 1 to Day 14 (0 [predose] to 15 hours postdose); Day 15 (24 hours post the Day 14 dose and before dosing on Day 15); and Day 16
Oral Clearance (CL/F) of Lu AF28996 | Day 1 to Day 14 (0 [predose] to 15 hours postdose); Day 15 (24 hours post the Day 14 dose and before dosing on Day 15); and Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Ehime University Hospital, Ehime, Japan